CLINICAL TRIAL: NCT01535924
Title: A Phase I/II Study Of Gemcitabine And Bendamustine In Patients With Relapsed Or Refractory Hodgkin's Lymphoma
Brief Title: Gemcitabine and Bendamustine in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Christian (Other)
Responsible Party: Sponsor-Investigator, Beth Christian, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-11015; NCI-2012-00022 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-06; First posted 2012-02-20 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Lymphocyte Predominant Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Recurrent Adult Hodgkin Lymphoma
Keywords: Hodgkin's Lymphoma; relapsed; refractory
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Gemcitabine; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1 and 2. Treatment repeats every 21-28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: bendamustine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda

SUMMARY:
This phase I/II trial studies the side effects and best dose of bendamustine hydrochloride when given together with gemcitabine hydrochloride and to see how well it works in treating patients with relapsed or refractory Hodgkin lymphoma. Drugs used in chemotherapy, such as gemcitabine hydrochloride and bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug, combination chemotherapy, may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity and determine the maximum tolerated dose (MTD) of combined bendamustine (bendamustine hydrochloride) and gemcitabine (gemcitabine hydrochloride) in patients with relapsed or refractory Hodgkin's lymphoma.

II. To determine the overall response rate of bendamustine and gemcitabine in patients with relapsed and refractory Hodgkin's lymphoma.

SECONDARY OBJECTIVES:

I. To determine whether therapy with bendamustine in the setting of relapsed or refractory Hodgkin's lymphoma will impact future stem cell collection.

OUTLINE: This is a phase I, dose-escalation study of bendamustine hydrochloride followed by a phase II study.

Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1 and 2. Treatment repeats every 21-28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 2 years, then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented Classical Hodgkin's lymphoma that is recurrent or refractory after standard chemotherapy; core biopsies are acceptable if they contain adequate tissue for primary diagnosis and immunophenotyping; bone marrow biopsies as the sole means of diagnosis are not acceptable
* Patients with Hodgkin's lymphoma may have one of the following World Health Organization subtypes:

  * Nodular sclerosis Hodgkin's lymphoma
  * Lymphocyte-rich Hodgkin's lymphoma
  * Mixed cellularity Hodgkin's lymphoma
  * Lymphocyte depletion Hodgkin's lymphoma
  * Nodular lymphocyte predominant Hodgkin's lymphoma
* Patients must have relapsed or progressed after at least one prior therapy
* Patients with relapsed or refractory disease following stem cell transplantation are permitted
* No prior treatment with bendamustine; prior therapy with gemcitabine is permitted
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable
* Measurable disease: lesions that can be accurately measured in at least two dimensions as >= 1.0 x 1.0 cm by computerized tomography (CT), PET/CT (positron emission tomography/CT), or magnetic resonance imaging (MRI)
* Non-measurable disease: all other lesions, including small lesions (less than 1.0 x 1.0 cm) and truly non-measurable lesions; lesions that are considered non-measurable include the following:

  * Bone lesions (lesions if present should be noted)
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonis
  * Bone marrow (involvement by Hodgkin's lymphoma should be noted)
* Non-pregnant and non-nursing; due to the teratogenic potential of these agents, pregnant or nursing patients may not be enrolled; women and men of reproductive potential should agree to use an effective means of birth control
* Patients with human immunodeficiency virus (HIV) infection are eligible; patients with HIV infection must meet the following: No evidence of co-infection with hepatitis B or C; cluster of differentiation (CD)4+ count >= 400/mm; no evidence of resistant strains of HIV; on anti-HIV therapy with an HIV viral load < 50 copies HIV ribonucleic acid (RNA)/mL; no history of acquired immune deficiency syndrome (AIDS) defining conditions

  * Granulocytes >= 1000/μl
  * Platelet count >= 75,000/μl
  * Creatinine =< 20 mg/dL
  * Bilirubin =< 2.0 mg/dL
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.0 x upper limits of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Christian, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Background] Cohen JB, Wei L, Maddocks KJ, Christian B, Heffner LT, Langston AA, Lechowicz MJ, Porcu P, Flowers CR, Devine SM, Blum KA. Gemcitabine and bendamustine is a safe and effective salvage regimen for patients with recurrent/refractory Hodgkin lymphoma: Results of a phase 1/2 study. Cancer. 2020 Mar 15;126(6):1235-1242. doi: 10.1002/cncr.32640. Epub 2019 Dec 10. PMID 31821549
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The current study was conducted at the Ohio State University in Columbus, Ohio, and Emory University in Atlanta, Georgia.
Groups:
- Phase 1 (Dose Level 1): Dose Level 1: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 60 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 1 (Dose Level 2): Dose Level 2: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 90 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 1 (Dose Level 3): Dose Level 3: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 120 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 1 (Dose Level 4): Dose Level 4: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 90 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 2 (Dose Level 5); Phase 2: Patients receive Gemcitabine 1000mg/m2 on day 1 and Bendamustine 120mg/m2 on days 1 and 2 of each 21 day cycle. Gemcitabine shall be administered prior to Bendamustine on day 1 of each cycle.
Period: Overall Study
Arm/Group | Phase 1 (Dose Level 1) | Phase 1 (Dose Level 2) | Phase 1 (Dose Level 3) | Phase 1 (Dose Level 4) | Phase 2 (Dose Level 5) | Phase 2
Started | 3 | 3 | 3 | 4 | 6 | 7
Completed | 3 | 3 | 3 | 4 | 6 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 (Dose Levels 1): Dose Level 1: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 60 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  gemcitabine hydrochloride: Given IV bendamustine hydrochloride: Given IV
- Phase 1 (Dose Levels 2): Dose Level 2: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 90 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 1 (Dose Levels 3): Dose Level 3: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 120 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 1 (Dose Levels 4): Dose Level 4: Patients receive Gemcitabine 1000 mg/m2 IV over 30 minutes on day 1 and Bendamustine 90 mg/m2 IV over 30 minutes on days 1 and 2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
- Phase 2 (Dose Levels 5); Phase 2: Patients receive Gemcitabine 1000mg/m2 on day 1 and Bendamustine 120mg/m2 on days 1 and 2 of each 21 day cycle. Gemcitabine shall be administered prior to Bendamustine on day 1 of each cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Dose Levels 1) | Phase 1 (Dose Levels 2) | Phase 1 (Dose Levels 3) | Phase 1 (Dose Levels 4) | Phase 2 (Dose Levels 5) | Phase 2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (17.34) | 38 (9.16) | 35 (11.63) | 50 (7.78) | 33.33 (16.05) | 37.14 (12.03) | 38.19 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 1 | 3 | 2 | 10
  Male | 2 | 2 | 1 | 3 | 3 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 4 | 6 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 1 | 3
  White | 3 | 2 | 1 | 4 | 5 | 6 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: patients]
  United States | 3 | 3 | 3 | 4 | 6 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events in Terms of Dose-limiting Toxicity (DLT) and MTD of Bendamustine Hydrochloride (Phase I)
Description: Dose limiting toxicity will be defined during cycle 1 only of the phase I trial. Hematologic and Infectious Dose Limiting Toxicities include: Grade 3 febrile neutropenia persisting> 7 days, Grade 4 infection or febrile neutropenia. Treatment delay>14 days due to grade 3-4 neutropenia or thrombocytopenia. Non-Hematological Dose Limiting Toxicities include: any Grade 3 or 4 non-hematologic toxicity related to study treatment with the exception of nausea or vomiting, alopecia, or electrolyte/glucose abnormalities that are correctable within 72 hours.
Time Frame: up to 5 years
Population: Only patients in Phase I analyzed
Measure: Number; unit: number of patients
Arm/Group | Phase 1 (Dose Levels 1) | Phase 1 (Dose Levels 2) | Phase 1 (Dose Levels 3) | Phase 1 (Dose Levels 4) | Phase 2 (Dose Levels 5) | Phase 2
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 0 | 0
number of patients | 0 | 0 | 0 | 0 |  |

2. Secondary Outcome: Overall Response Rate (ORR) of Bendamustine Hydrochloride and Gemcitabine Hydrochloride in Patients With Relapsed or Refractory Hodgkin Lymphoma (Phase II)
Description: Tested using Simon's two-stage Minimax design. Descriptive statistics (i.e. means, standard deviations, 95% confidence intervals for continuous variables, and frequencies for discrete data) and graphical analyses will be used for all correlative laboratory parameters. The associations between correlative laboratory parameters and clinical response will be evaluated using two sample t test or Fisher's exact test, whichever is appropriate.
Time Frame: up to 5 years
Population: Only patients in Phase II analyzed
Measure: Number; unit: percentage of patients
Arm/Group | Phase 1 (Dose Levels 1) | Phase 1 (Dose Levels 2) | Phase 1 (Dose Levels 3) | Phase 1 (Dose Levels 4) | Phase 2 (Dose Levels 5) | Phase 2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 6 | 7
percentage of patients |  |  |  |  | 67 | 71

ADVERSE EVENTS:
Time Frame: The Adverse event information was collected for study patients from baseline through study completion utilizing the CTCAE version 4.0 to determine the severity of the reaction for adverse event reporting from baseline to after study completion, up to 5 years.
Description: The National Cancer Institutes Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Arm/Group | Phase 1 (Dose Levels 1) | Phase 1 (Dose Levels 2) | Phase 1 (Dose Levels 3) | Phase 1 (Dose Levels 4) | Phase 2 (Dose Levels 5) | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/4 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 0/3 | 4/4 | 1/6 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Dose Levels 1) (N=3) | Phase 1 (Dose Levels 2) (N=3) | Phase 1 (Dose Levels 3) (N=3) | Phase 1 (Dose Levels 4) (N=4) | Phase 2 (Dose Levels 5) (N=6) | Phase 2 (N=7)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune Systems Disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection and Infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraoperative urinary injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Dose Levels 1) (N=3) | Phase 1 (Dose Levels 2) (N=3) | Phase 1 (Dose Levels 3) (N=3) | Phase 1 (Dose Levels 4) (N=4) | Phase 2 (Dose Levels 5) (N=6) | Phase 2 (N=7)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 1 (2) | 2 (2) | 3 (5) | 2 (4)
Alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (5) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 2 (4) | 3 (3) | 2 (2) | 6 (7) | 7 (9)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Fever (General disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 3 (3)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 2 (3) | 3 (3) | 2 (2) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 3 (5) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Lung infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 3 (9) | 3 (4) | 4 (4) | 6 (7) | 7 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (11) | 2 (4) | 4 (6) | 4 (5) | 5 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (3) | 1 (4) | 2 (3) | 4 (5) | 3 (6) | 4 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (2) | 2 (5) | 3 (6) | 2 (2)
White blood cell decreased (Investigations) | 2 (2) | 1 (1) | 3 (5) | 1 (1) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 0 (0) | 2 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT01535924/Prot_SAP_000.pdf